CLINICAL TRIAL: NCT03894839
Title: Evaluation of the Effect of Different Cleaning and Disinfection Procedures on the Involvement of Candida Species
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Beyza Ünalan Değirmenci, Assistant Professor, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20.06.2017/01
Record Dates: First submitted 2019-03-18; First posted 2019-03-29 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Candidiasis, Oral
Keywords: Prothesis stomatitis, disinfection methods
MeSH Terms: conditions — Candidiasis, Oral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- glutaraldehyde disinfection and microwave application (Active Comparator): %2 glutaraldehyde, solution form,duration time 1 minute and 1 time in a day by patients and 3 minutes 650 watt microwave energy application by dentists at each control session
  Interventions: Other: glutaraldehyde disinfection and microwave application
- Chlorhexidine gluconate disinfection and microwave application (Active Comparator): %2 chlorhexidine gluconate, solution form, duration time 1 minute and 1 time in a day by patients and 3 minutes 650 watt microwave energy application by dentists at each control session
  Interventions: Other: Chlorhexidine gluconate disinfection and microwave application
- Sodium hypochlorite disinfection and microwave application (Active Comparator): %5 sodium hypochlorite, solution form,duration time 1 minute and 1 time in a day by patients and 3 minutes 650 watt microwave energy application by dentists at each control session
  Interventions: Other: Sodium hypochlorite disinfection and microwave application
- glutaraldehyde disinfection and ozone therapy (Active Comparator): %2 glutaraldehyde, solution form,duration time 1 minute and 1 time in a day by patients and 15 minutes ozone therapy at each control session by dentists
  Interventions: Other: glutaraldehyde disinfection and ozone therapy
- Chlorhexidine gluconate disinfection and ozone therapy (Active Comparator): %2 chlorhexidine gluconate, solution form, duration time 1 minute and 1 time in a day by patients and 15 minutes ozone therapy at each control session by dentists
  Interventions: Other: Chlorhexidine gluconate disinfection and ozone therapy
- Sodium hypochlorite disinfection and ozone therapy (Active Comparator): %5 sodium hypochlorite, solution form,duration time 1 minute and 1 time in a day by patients and 15 minutes ozone therapy at each control session by dentists
  Interventions: Other: Sodium hypochlorite disinfection and ozone therapy

INTERVENTIONS:
Other: glutaraldehyde disinfection and microwave application — Combination of the chemical disinfection which could be done by patients and professional disinfection methods which is done by dentists
  Arms: glutaraldehyde disinfection and microwave application
Other: Chlorhexidine gluconate disinfection and microwave application — Combination of the chemical disinfection which could be done by patients and professional disinfection methods which is done by dentists
  Arms: Chlorhexidine gluconate disinfection and microwave application
Other: Sodium hypochlorite disinfection and microwave application — Combination of the chemical disinfection which could be done by patients and professional disinfection methods which is done by dentists
  Arms: Sodium hypochlorite disinfection and microwave application
Other: glutaraldehyde disinfection and ozone therapy — Combination of the chemical disinfection which could be done by patients and professional disinfection methods which is done by dentists
  Arms: glutaraldehyde disinfection and ozone therapy
Other: Chlorhexidine gluconate disinfection and ozone therapy — Combination of the chemical disinfection which could be done by patients and professional disinfection methods which is done by dentists
  Arms: Chlorhexidine gluconate disinfection and ozone therapy
Other: Sodium hypochlorite disinfection and ozone therapy — Combination of the chemical disinfection which could be done by patients and professional disinfection methods which is done by dentists
  Arms: Sodium hypochlorite disinfection and ozone therapy

SUMMARY:
Individuals may experience tooth loss as a result of trauma, periodontal destruction, lack of adequate bone support and clinically dental mobility. The increase in these tooth loss results in a condition called complete toothlessness in patients, and as a result of this, dentists treat complete dentures. It is known that the microorganism retention in the existing restorations is faster and higher than the natural tissues, and this leads to faster plaque build-up and hence bad odor. Candida species are common in oral flora, because they are numerous in the mouth and they are opportunistic pathogenic fungi that can make superficial and deep infections. The most important pathogen species among these parasites is Candida albicans. Mouth moniliasis or acute pseudomembrane candidiasis in the oral cavity of the so-called canker is caused by C.albicans. Chronic hyperplastic candidiasis is a clinical entity that is clinically inseparable from leukoplakia and completely separate from thrush. The accumulation of microorganisms in prosthetic materials is very important for the protection of the health of oral tissues and it is desirable to use appropriate cleaning and disinfection materials to minimize this accumulation.

It is known in the literature that ozone and microwave technologies are used as disinfection technique. In this study, the application of ozone and microwave technologies in addition to the cleaning agents used as standard treatment will be compared in vivo. No such research has been found.The aim of this study was to evaluate the effect of different cleaning and disinfection procedures on the involvement of Candida species in complete denture patients.

DETAILED DESCRIPTION:
The study is planned to be performed on 72 patients between the ages of 18-70 who were diagnosed and followed up in the Department of Prosthodontics of the Faculty of Dentistry of Yuzuncu Yil University. Patients with complete disability and indication of total prosthesis are included in the case group. In addition, individuals with systemic disturbance of salivation, radiotherapy-chemotherapy patients who are known to be able to facilitate Candida growth will be excluded from our study. The complete prosthesis made of polymethylmethacrylate material will be delivered to the patients. Before delivery, the polished surfaces of the relevant prosthesis, its vertical size, whether the patient is suitable for use or not, and the delivery of the prostheses that have passed the relevant controls will be considered appropriate. Patients will be asked to come for follow-up at 1 week and 1 month after the delivery of full dentures. The patients will be delivered with one of the glutaraldehyde, sodium hypochlorite or chlorhexidine digluconate solutions as the cleaning solution determined by the researchers during the initial delivery of their prostheses. Patients will be asked to clean with this relevant solution twice a day, in accordance with the specified times. At the 1 st and 1 st month follow-up, the prosthesis will be taken for the determination of the Candida number and species and the following procedures will be applied. Delivered prostheses will be taken in a 250 ml beaker (containing 100 ml of distilled water). Then, with the help of a swab, it will be contacted to the inner surfaces and edges of the prosthesis to allow mixing into the distilled water in possible biofilm layers.

Then, the prosthesis will be removed and the distilled water will be homogenized by mixing thoroughly with the help of a stirrer. Later Zhou et al. According to the method used; 1 ml of distilled water will be transferred to falcon tubes. Pre-cultural Falcon tubes will be kept on ice for up to 1 hour.

Prior to culture, samples will be diluted with sterile distilled water (1: 1, 1:10, 1: 100). And be mixed well using a vortex mixer. Then take 0.5 ml of these diluted liquids to be planted in Sabouraud Dextrose Agar. After 48 hours of incubation (microscopic and macroscopic evaluation), the number of colony forming units (CFU) of distilled water will be counted using two researchers. Then, Candida lara will be identified by an API test which will include 19 carbohydrate assimilation tests and negative control.

The same processes will be repeated after the disinfection process with ozone or microwave to compare the effectiveness of the disinfection process. Thus, the daily recommended by physicians for the daily cleaning process, the suppression of reproduction and reproduction of Candida species, and a new method proposed by physicians to be applied as a new method of ozone and microwave and how much efficiency of sterilization on the Candida number will be compared on the basis of the effects will be compared.

Statistical analysis will be done and interpreted.

ELIGIBILITY:
Inclusion Criteria:

* Patients without any teeth
* Patients who had indicated to doing denture

Exclusion Criteria:

* patients with hyposalivation
* patients who use the medication that affects salivation
* patients who have chemotherapy or radiotherapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2018-10-26 (Actual); Study Completion 2019-01-22 (Actual)

PRIMARY OUTCOMES:
Numbers and the types of Candida species that isolated from denture base after daily used disinfections on at 1st week | 1 week
  Chemical disinfectants which were used by patients must decreased the number of Candida species that eliminated from denture surfaces.
Numbers and the types of Candida species that isolated from denture base after professionally used disinfection methods on at 1st week | 1 week
  Disinfection methods which were done by dentists must decreased the number of Candida species that eliminated from denture surfaces.
Numbers and the types of Candida species that isolated from denture base after daily used disinfections on at 1st month | 1 month
  Chemical disinfectants which were used by patients must decreased the number of Candida species that eliminated from denture surfaces.
Numbers and the types of Candida species that isolated from denture base after professionally used disinfection methods on at 1st month | 1 month
  Chemical disinfectants which were used by patients must decreased the number of Candida species that eliminated from denture surfaces.

CONTACTS AND LOCATIONS:
Locations (1):
- Beyza Ünalan Değirmenci, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mojarad N, Khalili Z, Aalaei S. A comparison of the efficacy of mechanical, chemical, and microwave radiation methods in disinfecting complete dentures. Dent Res J (Isfahan). 2017 Mar-Apr;14(2):131-136. PMID 28584537
- [Result] Pires CW, Fraga S, Beck AC, Braun KO, Peres PE. Chemical Methods for Cleaning Conventional Dentures: What is the Best Antimicrobial Option? An In Vitro Study. Oral Health Prev Dent. 2017;15(1):73-77. doi: 10.3290/j.ohpd.a37716. PMID 28232977
- [Result] Aslanimehr M, Mojarad N, Ranjbar S, Aalaei S. In vitro comparison of the effects of microwave irradiation and chemical and mechanical methods on the disinfection of complete dentures contaminated with Candida albicans. Dent Res J (Isfahan). 2018 Sep-Oct;15(5):340-346. PMID 30233654